CLINICAL TRIAL: NCT04151888
Title: Evaluation of Nasal Hot Water Irrigation in the Management of Posterior Epistaxis
Brief Title: Hot Water Irrigation in Posterior Epistaxis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RT Fahmy, Resident doctor, Assiut University
Other Study IDs: Epistaxis
Record Dates: First submitted 2019-10-18; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Foley catheter — Thin sterile tube will be inserted in choana

SUMMARY:
This study was aimed to assess the efficacy and factors affecting the success of hot water irrigation in management of posterior epistaxis.

DETAILED DESCRIPTION:
Epistaxis has been reported to occur in up to 60% of general population.This condition has incidence peaks at ages younger than 10 years and older than 50 years. Epistaxis appears to occur more in males than females . In rare cases massive nasal bleeding can lead to death.

Nasal bleeding usually responds to first aid measures such as compression.When Epistaxis doesn't respond to simple measures. The source of bleeding should be located and treated appropriately. Treatment options to be considered include topical vasoconstriction, chemical cautery, electrocautery, nasal packing, posterior gauze packing, use of balloon system, and arterial ligation or embolization. Hospital admission should be considered with patients with comorbid conditions or complication of blood loss.

Nasal Hot water irrigation was first described by Guice in 1878 as an effective method of treating severe life-threatening epistaxis. However, the technique was already in use by nineteenth century obstetricians as a method of treating postpartum bleeding . In the second half of the twenties century, nasal packing products and the development of endoscopic sinus surgery almost completely replaced the irrigation technique as treatment for posterior epistaxis. However, Stangerup et al. (1996) have demonstrated that hot water irrigation, using temperatures of up to 50°C, produces vasodilation and oedema of the nasal mucosa without the risk of necrosis and accelerating the clotting cascade.

Hot water irrigation had a higher success rate (55 %) in treating posterior epistaxis, compared with nasal packing (44 %) .Using a modified irrigation technique, was able to stop bleeding permanently in up to 82 %of cases of posterior epistaxis, including patients receiving antiplatelet agents or anticoagulants . During a follow-up period of four to 24 months. Furthermore, successful hot water irrigation was associated with less nasal trauma, significantly less pain, fewer surgical procedures and avoidance of a hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* patients age: > 10 years.
* Failed first aid measures.

Exclusion Criteria:

* Patients age < 10 years old.
* Patients with anterior epistaxis.
* Patients presented with hemorrhagic shock.
* Patients presented with post-surgical bleeding.
* Suspected nasal pathology e.g tumors or trauma.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is including patients with spontaneous posterior epistaxis referred to ENT Department, Assiut University Hospital. .
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-30 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of hot water irrigation in management of posterior epistaxis | 2 years
  Observation of the patients for 24 hrs after controlling of posterior epistaxis using hot water irrigation if it can control posterior epistaxis or not and this will be confirmed by using coagulation profile and complete blood count

REFERENCES:
- [Background] Randall DA, Freeman SB. Management of anterior and posterior epistaxis. Am Fam Physician. 1991 Jun;43(6):2007-14. PMID 2042544